CLINICAL TRIAL: NCT05651230
Title: Seaweed-derived Rhamnan Sulfate and Vascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: Konan Chemical Manufacturing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00003693
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhamnan sulfate (Experimental): The subjects will take rhamnan sulfate (Rhamnox100, Konan Chemical Manufacturing Co. LTD, Mie, Japan: 540 mg/day) orally three time daily at each meal time.
  Interventions: Dietary Supplement: Rhamnan sulfate
- Placebo (Placebo Comparator): The subjects will take placebo (Konan Chemical Manufacturing Co. LTD, Mie, Japan: 540 mg/day) orally three time daily at each meal time.
  Interventions: Dietary Supplement: Rhamnan sulfate

INTERVENTIONS:
Dietary Supplement: Rhamnan sulfate — A randomized, placebo-controlled, double-blind crossover dietary supplement intervention consisting of 3 weeks each of rhamnan sulfate (Rhamnox100, Konan Chemical Manufacturing Co. LTD, Mie, Japan: 540 mg/day) or placebo with 2 weeks of washout between the interventions will be conducted. Dietary supplements (rhamnan sulfate) will be taken orally three time daily at each meal time. Rhamnan sulfate is a polysaccharide (carbohydrate) extracted from seaweeds and can be considered nutrition supplement. As each pill contains 90 mg of rhamnan sulfate or placebo, subjects will be taking 2 pills before or during each meal.
  Other Names: Rhamnox100

SUMMARY:
The primary aim of the proposed investigation is to examine the hypothesis that a relatively short period of rhamnan sulfate supplementation would improve key markers of vascular dysfunction in middle-aged and older adults with at least one risk factors for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* at least one risk factor for cardiovascular disease (e.g., dyslipidemia, hypertension, obesity, impaired fasting glucose)
* a BMI of <40 kg/m2

Exclusion Criteria:

* gastrointestinal disorders and/or renal disease
* pregnancy or lactation
* strenuous physical activity (>3 times/week)
* alcohol abuse

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Vascular function | Before the 3-week intervention
  Endothelium-dependent vasodilation as assessed by flow-mediated dilation
Vascular function | After the 3-week intervention
  Endothelium-dependent vasodilation as assessed by flow-mediated dilation

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Aging Research Lab at UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request after the research findings are published.